CLINICAL TRIAL: NCT06291519
Title: The Effect of Multisensory Stimulus Method Used During Immunisation on Pain and Physiological Parameters in Infants: A Randomised Controlled Study
Brief Title: The Effect of Multisensory Stimulus Method on Pain and Physiological Parameters in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kadriye Sahin, Research Assistant -( RN, MSc, PhDc), Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SHN50343434
Record Dates: First submitted 2024-02-06; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Multisensory Stimulation
Keywords: Infant baby; Multisensory stimulation; newborns; vaccine; pain; nursing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group 1 (Experimental): In this group, the mother applied multiple sensory stimuli. In this group, the mothers of the babies to be vaccinated applied multiple sensory stimuli such as breastfeeding, mother's voice, touch-light massage, and eye contact. The mother breastfed her baby for a total of 20 minutes. Breastfeeding was terminated before vaccination. Other applications were applied for 5 minutes before vaccination and 5 minutes after vaccination. FLACC pain scale, SPO2, and pulse oximetry were evaluated and recorded 5 min before and 2 min after vaccination, immediately before vaccination, immediately after vaccination (pain during the procedure), and 2 and 5 min after the procedure.
  Interventions: Other: Multi-sensory Stimulation Method-Mother Applying the Method to the Baby
- Experimental Group 2 (Experimental): In this group, the nurse applied multiple sensory stimuli. In this group, the mothers of the babies to be vaccinated breastfed the baby for 20 minutes. The mother stopped breastfeeding before the vaccination procedure. The nurse started to give multisensory stimuli. The nurse administered multisensory stimuli including soft tone of voice, touch-light massage, and eye contact 5 minutes before the vaccination. Other applications were applied 5 minutes before and 5 minutes after vaccination. FLACC pain scale, SPO2, and pulse oximetry were evaluated and recorded 5 min before and 2 min after vaccination, immediately before vaccination, immediately after vaccination (pain during the procedure), and 2 and 5 min after the procedure.
  Interventions: Other: Multi-sensory Stimulation Method-Nurse Applying the Method to the Baby
- Experimental Group 3 (Experimental): In this group, the mother breastfed her baby for 20 minutes before vaccination. Breastfeeding was terminated before vaccination. FLACC pain scale, SPO2, and pulse oximetry were evaluated and recorded 5 min before and 2 min after vaccination, immediately before vaccination, immediately after vaccination (pain during the procedure), and 2 and 5 min after the procedure.
  Interventions: Other: Breastfeeding Applied Group
- Control Group (No Intervention): Babies in this group did not receive any treatment. A light touch was applied for ethical reasons. FLACC pain scale, SPO2, and pulse oximetry were evaluated and recorded 5 min before and 2 min after vaccination, immediately before vaccination, immediately after vaccination (pain during the procedure), and 2 and 5 min after the procedure.

INTERVENTIONS:
Other: Multi-sensory Stimulation Method-Mother Applying the Method to the Baby — In the multisensory stimulus method;
  1. st stimulus (sense of taste): The mother breastfed the baby for 20 minutes. Breastfeeding was terminated before vaccination.
  2. nd stimulus (sense of touch),: The mother applied touch - a light massage for 5 min until the vaccination process. There was a break just before the vaccination. The application was continued for another 5 min after the vaccination.
  3. rd stimulus: Speech-Sound (sense of hearing): The mother spoke to the baby in a soft tone for 5 minutes until the vaccination (words, lullabies, songs, etc.). There was a break just before the vaccination. The practice was continued for 5 minutes immediately after the vaccination.
  4. Stimulus Eye contact (sense of sight): The mother made eye contact with the baby in the mother's field of vision for 5 minutes until the vaccination. There was a break just before the vaccination. The application continued for another 5 minutes after the vaccination.
  Arms: Experimental Group 1
Other: Multi-sensory Stimulation Method-Nurse Applying the Method to the Baby — In the multisensory stimulus method;
  1. st stimulus (sense of taste): The mother breastfed the baby for 20 minutes. Breastfeeding was terminated 5 min before vaccination.
  2. nd stimulus (sense of touch),: The nurse applied touch - a light massage for 5 minutes until the vaccination. There was a break just before the vaccination. The application was continued for another 5 min after the vaccination.
  3. rd stimulus: Speech-Sound (sense of hearing): The nurse spoke to the baby in a soft tone for 5 minutes until the vaccination (words, lullabies, songs, etc.). There was a break just before the vaccination. The practice was continued for 5 minutes immediately after the vaccination.
  4. Stimulus Eye contact (sense of sight): The nurse made eye contact with the baby in the mother's field of vision for 5 minutes until the vaccination. There was a break just before the vaccination. The application continued for another 5 minutes after the vaccination.
  Arms: Experimental Group 2
Other: Breastfeeding Applied Group — Multisensory stimulus method not applied:
  The baby was breastfed by its mother for 20 minutes. Breastfeeding was stopped just before the vaccination.
  Arms: Experimental Group 3

SUMMARY:
This study aimed to investigate the impact of employing the multi-sensory stimulation technique by both the mother and the nurse on the pain and physiological responses of infants aged 2-6 months during vaccination. The significance of pain experienced during vaccination in children is emphasized, potentially leading to avoidance behaviors toward healthcare services. There is growing evidence supporting the efficacy of non-pharmacological interventions. Multi-sensory stimulation, which integrates various stimuli such as taste, touch, and speech, alleviates infant pain. However, there has been a lack of studies assessing the effectiveness of this approach during vaccination administered by different healthcare providers. Hence, this study sought to explore the effects of multi-sensory stimulation by both mother and nurse applied to pain and physiological parameters. It is anticipated that the findings of this study will contribute to both pain management strategies and healthcare practices.

DETAILED DESCRIPTION:
The emergence of needle phobia in childhood often precipitates avoidance behaviors toward vaccinations (McLenon & Rogers, 2019). Mitigating vaccine-induced pain holds promise in alleviating healthcare avoidance inclinations (Komaroff & Forest, 2020). An expanding body of evidence substantiates the efficacy of non-pharmacological interventions in ameliorating acute procedural pain in neonates and infants (Aydın & İnal, 2019; Reece-Stremtan & Gray, 2016).

One such auspicious non-pharmacological approach to pain management is multisensory stimulation, also recognized as sensory saturation. Multisensory stimulation constitutes a non-pharmacological strategy employed to diminish infant pain during acute procedures. Grounded in gate control theory, it postulates that administering both a sweet taste and a spectrum of stimuli to infants may yield heightened analgesic effects (Bellini et al., 2012). The amalgamation of various interventions such as massage, auditory stimuli, olfactory cues, and eye contact via multisensory stimulation engages broader cortical regions and saturates sensory pathways, thereby attenuating nociceptive inputs (Zeraati et al., 2017).

A review of the literature underscores the efficacy of multisensory stimulation as a non-pharmacological modality to alleviate painful procedures in preterm neonates (Anand et al., 2011). Moreover, it demonstrates superior efficacy compared to single pain relief modalities in mitigating pain during venipuncture in infants (Fitri et al., 2020). Despite the demonstrated efficacy of multisensory stimulation as a straightforward, effective, and safe analgesic method during painful neonatal examinations, studies evaluating its effectiveness during vaccine administration are notably absent. Furthermore, scant research has explored the influence of the practitioner (whether mother, nurse, or physician) on the efficacy of this method.

Hypotheses : Babies who underwent the multi-sensory stimulation method; the Pain scale score is lower than the control group, the crying duration is shorter than the control group, the heart rate is lower than the control group, and the saturation (SPO2) is higher than the control group. In the group where the mother is the practitioner of the Multi-sensory stimulation method, compared to the group where the nurse is the practitioner; the pain scale score is low, the crying duration is low, the heart rate is low, saturation level (SPO2) is high.

Aim:

Hence, this study aims to investigate the impact of multisensory stimulation administered by both mothers and nurses on pain perception and physiological parameters during vaccine administration.

Place and Time of the Research:

The data were collected at the Healthy Child Vaccination Unit of a university hospital by visiting the institution two days a week, on Thursdays and Fridays, between January 2023 and December 2023.

Universe and Sample After obtaining the necessary legal permissions (ethics committee approval and institutional permission), the population of the study consisted of infants between the ages of 2-6 months who were applied to the Istanbul University Cerrahpaşa Medical Faculty vaccination room by their mothers for routine vaccination on the dates of the study.

The research sample consisted of 96 infants between the ages of 2-6 months who were brought to the vaccination room between January 2023 and October 2023, met the inclusion criteria, and whose parents gave written informed consent. According to the power analysis, a total of 96 babies were kept safe, 24 babies per group.

Randomization Babies who met the research selection criteria were the group in which the multi-sensory stimulation method was applied, the approved group of the multi-sensory stimulation method, the experimental group, the breastfeeding group, and the control group according to age (2 months, 4 months, 6 months) in which the block randomization method was mostly applied.

Independent variables: Multi-sensory stimulation method Dependent variables: Duration of infant crying, FLACC pain scale score, peak heart rate, saturation (SPO2) level.

Data Collection Method The data were collected by the researcher in the unit where the research was conducted

Data Collection Tools

* Data Collection Form prepared by the researcher to determine the demographic characteristics of the baby. Some information (such as gestational week, gender, and anthropometric measurements at birth) was obtained from the child's personal records.
* FLACC scale to determine the pain score before, during, and after vaccination of infants,
* Pulse Oximetry Device to detect oxygen saturation (SPO2) and heart rate before, during and after immunization of infants,
* Weighing Instrument for determining the current weight of infants,
* Height Measuring Tape for determining the current height of babies,
* Multi-sensory stimulation method

Procedure The babies included in the study were divided into 4 groups by block randomization method after obtaining ethical and institutional permission. Multi-sensory stimulation method was applied by the mother to the 1st experimental group and by the nurse to the 2nd experimental group. In the breastfeeding group, the mother only breastfed, and no application was applied to the control group.

In all groups, FLACC pain scale, oxygen saturation, and pulse oximetry were evaluated and recorded 5 minutes and 2 minutes before the vaccination process, just before the vaccination, immediately after the vaccination (pain during the procedure), and at the 2nd and 5th minutes after the procedure. Post-vaccination crying duration was recorded in all groups.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Parental consent to participate in the study
* Born between 38-42 weeks of gestation
* To take part in the routine vaccination programme of the Ministry of Health

Exclusion Criteria:

* - Having taken analgesic, muscle relaxant or sedation within the last 4 hours

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
The Effect of Multiple Sensory Stimulus Method | Measured 5 minutes before, 2 minutes before, immediately before, immediately after, 2 minutes after and 5 minutes after vaccination in all groups
  The FLACC pain scale score decreased, the oxygen saturation value measured by pulse oximetry was measured higher, the heart rate measured by pulse oximetry was measured lower, and the crying time measured by stopwatch was measured lower in the infants who underwent multisensory stimulus method compared to the control group.

SECONDARY OUTCOMES:
Comparison of the group in which the mother applied multiple sensory stimuli and the group in which the nurse applied multiple sensory stimuli | Measured 5 minutes before, 2 minutes before, immediately before, immediately after, 2 minutes after and 5 minutes after vaccination in all groups
  The pain score measured with the FLACC pain scale was lower, the oxygen saturation value measured with pulse pulse oximetry was higher, there was no statistically significant difference between the heart rate values, and the crying time measured with a stopwatch was less in the group in which the mother applied multiple sensory stimuli during the vaccination procedure compared to the nurse group.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Yıldız, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, None Selected, Turkey (Türkiye)

REFERENCES:
- [Result] McLenon J, Rogers MAM. The fear of needles: A systematic review and meta-analysis. J Adv Nurs. 2019 Jan;75(1):30-42. doi: 10.1111/jan.13818. Epub 2018 Sep 11. PMID 30109720
- [Result] Komaroff A, Forest S. Implementing a clinical protocol using breastfeeding to mitigate vaccination pain in infants. J Pediatr Nurs. 2020 Sep-Oct;54:50-57. doi: 10.1016/j.pedn.2020.05.017. Epub 2020 Jun 10. PMID 32534408
- [Result] Aydin D, Inal S. Effects of breastfeeding and heel warming on pain levels during heel stick in neonates. Int J Nurs Pract. 2019 Jun;25(3):e12734. doi: 10.1111/ijn.12734. Epub 2019 Apr 17. PMID 30993840
- [Result] Reece-Stremtan S, Gray L. ABM Clinical Protocol #23: Nonpharmacological Management of Procedure-Related Pain in the Breastfeeding Infant, Revised 2016. Breastfeed Med. 2016 Nov;11:425-429. doi: 10.1089/bfm.2016.29025.srs. Epub 2016 Sep 13. PMID 27623411
- [Result] Bellieni CV, Tei M, Coccina F, Buonocore G. Sensorial saturation for infants' pain. J Matern Fetal Neonatal Med. 2012 Apr;25 Suppl 1:79-81. doi: 10.3109/14767058.2012.663548. Epub 2012 Mar 7. PMID 22339420
- [Result] Zeraati H, Shahinfar J, Behnam Vashani H, Reyhani T. Effect of Multisensory Stimulation on Pain of Eye Examination in Preterm Infants. Anesth Pain Med. 2016 Dec 7;7(1):e42561. doi: 10.5812/aapm.42561. eCollection 2017 Feb. PMID 28920044
- [Result] Anand KJS, Berqvist L, Hall RW, Carbajal R. (2011). Acute pain management in newborn infants. Pain:Clin Updat.;19(6):1 -6. 11 .
- [Result] Fitri SYR, Lusmilasari L, Juffrie M, Bellieni CV. Modified Sensory Stimulation Using Breastmilk for Reducing Pain Intensity in Neonates in Indonesia: A Randomized Controlled Trial. J Pediatr Nurs. 2020 Jul-Aug;53:e199-e203. doi: 10.1016/j.pedn.2020.04.004. Epub 2020 May 10. PMID 32402558
- [Derived] Sahin K, Yildiz S, Gur E. The effect of multi-sensory stimuli used during vaccination on pain and physiological parameters in infants: A randomized controlled trial. J Pediatr Nurs. 2026 Jan 6;87:20-30. doi: 10.1016/j.pedn.2025.11.051. Online ahead of print. PMID 41500000